CLINICAL TRIAL: NCT00004067
Title: A Randomized Trial Comparing the Safety and Efficacy of Adriamycin and Cyclophosphamide Followed by Taxol (AC-T) to That of Adriamycin and Cyclophosphamide Followed by Taxol Plus Herceptin (AC-T+H) in Node-Positive Breast Cancer Patients Who Have Tumors That Overexpress HER2
Brief Title: Doxorubicin and Cyclophosphamide Plus Paclitaxel With or Without Trastuzumab in Treating Women With Node-Positive Breast Cancer That Overexpresses HER2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP B-31; CDR0000067269
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Doxorubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: adriamycin + cyclophosphamide then taxol (Active Comparator)
  Interventions: Drug: adriamycin; Drug: cyclophosphamide; Drug: taxol
- Arm 2: adriamycin + cyclophosphamide then taxol + herceptin (Experimental)
  Interventions: Biological: herceptin; Drug: adriamycin; Drug: cyclophosphamide; Drug: taxol

INTERVENTIONS:
Biological: herceptin — 4 mg/kg loading dose then 2 mg/kg weekly for 1 year.
  Other Names: trastuzumab
  Arms: Arm 2: adriamycin + cyclophosphamide then taxol + herceptin
Drug: adriamycin — 60 mg/m2 IV push every 21 days for 4 cycles.
  Other Names: doxorubicin
Drug: cyclophosphamide — 600 mg/m2 IV every 21 days for 4 cycles
Drug: taxol — 175 mg/m2 IV every 21 days for 4 cycles
  Other Names: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin, cyclophosphamide, and paclitaxel, use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. It is not yet known whether combination chemotherapy plus trastuzumab is more effective than combination chemotherapy alone for treating breast cancer.

PURPOSE: This randomized phase III trial is studying how well giving combination chemotherapy together with trastuzumab works compared to combination chemotherapy alone in treating women with node-positive stage II or stage IIIA breast cancer that overexpresses HER2.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the cardiotoxicity of doxorubicin and cyclophosphamide followed by paclitaxel with or without trastuzumab (Herceptin®) in women with operable, node-positive breast cancer that overexpresses HER2.
* Compare the effect of these regimens on disease-free and overall survival of these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to number of positive nodes (1-3 vs 4-9 vs 10 or more), administration of hormonal therapy (tamoxifen vs anastrozole vs neither), surgery/radiotherapy (lumpectomy plus breast irradiation vs lumpectomy plus breast irradiation plus regional irradiation vs mastectomy without radiotherapy vs mastectomy with radiotherapy), paclitaxel schedule (every 3 weeks vs weekly), and participating center. Patients are randomized to one of two treatment arms.

* Arm 1: Patients receive doxorubicin IV and cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 21 days for 4 courses. Approximately 3 weeks after the last course, patients receive paclitaxel IV over 3 hours every 21 days for 4 courses OR paclitaxel IV over 1 hour once weekly for 12 weeks (12 doses).
* Arm 2: Patients receive chemotherapy as in arm I and trastuzumab (Herceptin®) IV over 90 minutes on day 1 of the first course of paclitaxel. Trastuzumab is then administered IV over 30 minutes weekly for 51 weeks, beginning on day 8.

All patients with estrogen or progesterone receptor-positive tumors receive hormonal therapy* for at least 5 years, beginning within 3-12 weeks after the last dose of chemotherapy. Patients who have received prior tamoxifen for prevention may be treated with additional tamoxifen for no more than 5 years at the discretion of the principal investigator (PI).

NOTE: *Other hormonal therapeutic agents are allowed in sequence with or as an alternative to tamoxifen therapy.

All patients previously treated with lumpectomy undergo breast irradiation beginning after completion of chemotherapy and concurrently with trastuzumab (in arm 2) administration. Patients previously treated with mastectomy may also receive radiotherapy. Radiotherapy is administered daily for 5-6 weeks.

Patients are followed every 6 months for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 2,700 patients will be accrued for this study within 4.75 years.

ELIGIBILITY:
Inclusion criteria

* The patient must have a life expectancy of at least 10 years, excluding her diagnosis of breast cancer. (Comorbid conditions should be taken into consideration, but not the diagnosis of breast cancer.)
* The interval between the last surgery for breast cancer treatment (lumpectomy, mastectomy, axillary dissection, or re-excision of lumpectomy margins) and randomization must be less than or equal to 84 days.
* All of the following staging criteria must be met:

  * Primary tumor must be T1-3 by clinical and pathologic evaluation.
  * Ipsilateral nodes must be cN0-1 by clinical evaluation.
  * Ipsilateral nodes must be pN1, pN2a, or pN3a by pathologic evaluation.
  * M0
* Patients must have undergone either a total mastectomy and an axillary dissection or a lumpectomy and an axillary dissection. Sentinel node biopsy is permitted, but must be followed by an axillary dissection.
* The tumor must be invasive adenocarcinoma on histologic examination.
* The tumor must be determined to be HER2-positive prior to randomization. Assays performed using fluorescent in situ hybridization (FISH) require gene amplification to be eligible. Assays using immunohistochemistry (IHC) must be performed at an NSABP-approved reference laboratory and require a strongly positive staining score.
* Patients must have an analysis of both estrogen and progesterone receptors performed on the primary tumor prior to randomization. "Marginal," "borderline," etc., results (i.e., those not definitely negative) will also be considered positive regardless of the methodology used.
* At the time of randomization, the patient must have had the following: history and physical exam, EKG, and PA and lateral chest x-ray within the past 3 months; and a bilateral mammogram (or unilateral if patient has had a mastectomy) and a pelvic exam (for women who have a uterus and who will be taking tamoxifen) within the past year.
* Within 3 months prior to entry, the patient must have a baseline left ventricular ejection fraction (LVEF) measured by MUGA scan equal to or greater than the lower limit of normal for the radiology facility. (If LVEF is > 75%, the investigator should consider having the LVEF determination reviewed prior to randomization. Following randomization, the LVEF determination may be reviewed up until the time of the post-AC MUGA. Please note that if a more accurate value is obtained from the review of the baseline MUGA, the corrected value must be submitted to the NSABP Biostatistical Center before the post-AC MUGA is performed.)
* At the time of randomization:

  * The postoperative absolute neutrophil count (ANC) must be ≥ 1500/mm3 (or <1500/mm3 if, in the opinion of the investigator, this represents an ethnic or racial variation of normal).
  * Postoperative platelet count must be ≥ 100,000/mm3. Significant underlying hematologic disorders must be excluded when the platelet count is above the upper limit of normal for the lab.
* There must be postoperative evidence of adequate hepatic function, i.e., total bilirubin must be ≤ ULN for the lab unless the patient has a chronic grade 1 bilirubin elevation (>ULN to ≤1.5 x ULN) due to Gilbert's disease or similar syndrome; and alkaline phosphatase must be <2.5 times the ULN for the lab; and the serum glutamic-oxaloacetic transaminase (SGOT [AST]) must be <1.5 times the ULN for the lab.
* There must be postoperative evidence of adequate renal function (serum creatinine within or less than the institution's normal range).
* Patients must have no clinical or radiologic evidence of metastatic disease. Suspicious findings must be confirmed as benign by radiologic evaluation or biopsy. A patient with skeletal pain is eligible for inclusion in the study if bone scan and/or roentgenological examination fails to disclose metastatic disease.
* Patients with a history of non-breast malignancies are eligible if they have been disease-free for 5 or more years prior to randomization and are deemed by their physician to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.
* Prior to randomization, the investigator must designate whether the patients who had a lumpectomy will receive local or locoregional radiation therapy. For patients who had a mastectomy, the investigator must designate whether or not the patient will receive radiation therapy. (Pre-randomization discussion and/or consultation with a radiation oncologist is encouraged.) Note: Irradiation of any internal mammary nodes is prohibited in this trial.
* Special conditions for eligibility of lumpectomy patients: irradiation and surgery
* Patients treated by lumpectomy and axillary node dissection to be followed by breast radiation therapy must meet all the eligibility criteria in addition to the following: Generally, lumpectomy should be reserved for tumors <5 cm. However, at the investigator's discretion, patients treated with lumpectomy for tumors ≥ 5 cm are eligible. The margins of the resected specimen must be histologically free of invasive tumor and DCIS as determined by the local pathologist. In patients in whom pathologic examination demonstrates tumor present at the line of resection, additional operative procedures may be performed to obtain clear margins. This is permissible even if axillary dissection has been performed. Patients in whom tumor is still present at the resected margin after re-excision(s) must undergo total mastectomy to be eligible. Whole breast irradiation is required. Irradiation of regional lymph nodes is optional, but partial breast irradiation and irradiation of any internal mammary nodes are prohibited in this trial. Intent to irradiate the axilla or other regional node groups must be declared by the investigator prior to randomization for stratification purposes.
* Special conditions for eligibility of mastectomy patients: irradiation. The decision to use locoregional irradiation in patients who have undergone total mastectomy and axillary node dissection must be declared by the investigator prior to randomization for stratification purposes. Failure to adhere to the radiation therapy plan will be a protocol violation.

Exclusion criteria

* Bilateral malignancy or a mass or mammographic abnormality in the opposite breast suspicious for malignancy unless there is biopsy proof that the mass is not malignant.
* Primary tumor staged as T4 for any reason.
* Nodes staged as clinical N2 or N3 for any reason and nodes staged as pathologic pN2b, pN3b, or pN3c.
* Prior history of breast cancer, including DCIS (patients with a history of lobular carcinoma in situ [LCIS] are eligible).
* Treatment including radiation therapy, chemotherapy, biotherapy, and/or hormonal therapy administered for the currently diagnosed breast cancer prior to randomization. The only exception is hormonal therapy, which may have been given for up to a total of 28 days anytime after diagnosis and before randomization. In such a case, hormonal therapy must stop at or before randomization and be re-started if indicated following chemotherapy.
* Prior anthracycline or taxane therapy for any malignancy.
* Any sex hormonal therapy, e.g., birth control pills, ovarian hormonal replacement therapy, etc. (These patients are eligible only if this therapy is discontinued prior to randomization.)
* Therapy with any hormonal agents such as raloxifene (Evista®), tamoxifen, or other selective estrogen receptor modulators (SERMs), either for osteoporosis or prevention. (Patients are eligible only if these medications are discontinued prior to randomization. These medications are not permitted while on the study except for the use of tamoxifen as described in the protocol)
* Nonmalignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude a patient from being subjected to any of the treatment options or would prevent prolonged follow-up.
* Cardiac disease that would preclude the use of Adriamycin, Taxol or Herceptin. This includes:
* Active cardiac disease:

  * angina pectoris that requires the use of antianginal medication;
  * cardiac arrhythmia requiring medication;
  * severe conduction abnormality;
  * clinically significant valvular disease;
  * cardiomegaly on chest x-ray;
  * ventricular hypertrophy on EKG; or
  * patients with poorly controlled hypertension, i.e., diastolic greater than 100 mm/Hg. (Patients with hypertension who are well controlled on medication are eligible for entry.)
* History of cardiac disease:

  * myocardial infarction documented as a clinical diagnosis or by EKG or any other tests;
  * documented congestive heart failure; or
  * documented cardiomyopathy.
* Psychiatric or addictive disorders that would preclude obtaining informed consent.
* Pregnancy or lactation at the time of proposed randomization. This protocol excludes pregnant or lactating women based on the fetal toxicity of both tamoxifen and Taxol which are listed as Pregnancy Category D agents. Pregnant women who received tamoxifen have experienced fetal deaths, birth defects, spontaneous abortions, and vaginal bleeding. Women of reproductive potential must agree to use an effective barrier method of contraception. Hormonal birth control methods are not permitted.
* Sensory/motor neuropathy ≥ grade 2, as defined by the NCI's Common Toxicity Criteria version 2.0.
* Contraindications to corticosteroid use which, in the opinion of the investigator, would preclude participation in this study.
* Concurrent treatment with other investigational agents.
* Sensitivity to benzyl alcohol.
* Special conditions for ineligibility of lumpectomy patients: irradiation and surgery. For patients treated by lumpectomy with axillary dissection, breast irradiation is required. Please see guidelines for radiation therapy in Appendix A. In addition, the following patients will also be ineligible:

  * Patients with diffuse tumors (as demonstrated on mammography) that would not be considered surgically amenable to lumpectomy.
  * Patients treated with lumpectomy in whom there is another clinically dominant mass or mammographically suspicious abnormality within the ipsilateral breast remnant. Such a mass must be biopsied and demonstrated to be histologically benign prior to randomization or, if malignant, must be surgically removed with clear margins.
  * Patients in whom the margins of the resected specimen are involved with invasive tumor or ductal carcinoma in situ (DCIS). Additional surgical resections to obtain free margins are allowed. Patients in whom tumor is still present after the additional resection(s) must undergo mastectomy to be eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2130 (Actual)
Dates: Start 2000-02; Primary Completion 2005-03 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | Time from randomization through 5 years
  Breast cancer recurrence, second primary cancer, death from any cause as first event
Cardiotoxicity | time from randomization through 4 months

SECONDARY OUTCOMES:
Survival | time from randomization through 5 years
  Death from any cause.
Long term effect of trastuzumab on cardiac function | At 5 and 10 years after randomization
  Ejection fraction will be measured by multigated acquisition scan (MUGA).

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (149):
- United States (141):
  - Comprehensive Cancer Institute, Huntsville, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Scripps Cancer Center at Scripps Clinic, La Jolla, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Pacific Shores Medical Group Comprehensive Hematology-Oncology Services - Long Beach, Long Beach, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Comprehensive Cancer Center at Desert Regional Medical Center, Palm Springs, California
  - Sutter Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Morton Plant Hospital, Clearwater, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - M.D. Anderson Cancer Center - Orlando, Orlando, Florida
  - Cancer Research Network, Inc., Plantation, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Rush Cancer Institute at Rush University Medical Center, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - West Suburban Hospital Medical Center, Oak Park, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Community Hospital, Munster, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Norton Cancer Center at Norton Hospital, Louisville, Kentucky
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Stanley S. Scott Cancer Center at Louisiana State University Medical Center - New Orleans, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Harry and Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - National Naval Medical Center, Bethesda, Maryland
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - New York Oncology Hematology, P.C. at Albany Regional Cancer Care, Albany, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Nalitt Cancer Institute at Staten Island University Hospital, Staten Island, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - Alamance Cancer Center, Burlington, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Leo W. Jenkins Cancer Center at Pitt County Memorial Hospital, Greenville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Akron City Hospital at Summa Health System, Akron, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Cancer Center at Jewish Hospital, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - South Pointe Hospital Cancer Care Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Cancer Care Center at Northside Medical Center, Youngstown, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - John and Dorothy Morgan Cancer Center at Lehigh Valley Hospital, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - York Cancer Center at Wellspan Health, York, Pennsylvania
  - Kent County Memorial Hospital, Warwick, Rhode Island
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Medical City Dallas Hospital, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - David Lee Cancer Center at Charleston Area Medical Center, Charleston, West Virginia
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Oncology Alliance, S.C. - Milwaukee, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Canada (8):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Carlo Fidani Peel Regional Cancer Centre at Credit Valley Hospital, Mississauga, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Royal Victoria Hospital - Montreal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec
  - Hopital du Saint-Sacrement, Quebec, Québec, Quebec

REFERENCES:
- [Background] Jahanzeb M. Adjuvant trastuzumab therapy for HER2-positive breast cancer. Clin Breast Cancer. 2008 Aug;8(4):324-33. doi: 10.3816/CBC.2008.n.037. PMID 18757259
- [Background] Reinholz MM, Dueck AC, Lingle WL, et al.: The concordance between NCCTG's and NSABP's C-myc FISH assays. [Abstract] J Clin Oncol 26 (Suppl 15): A-22110, 2008.
- [Background] Garrison LP Jr, Lubeck D, Lalla D, Paton V, Dueck A, Perez EA. Cost-effectiveness analysis of trastuzumab in the adjuvant setting for treatment of HER2-positive breast cancer. Cancer. 2007 Aug 1;110(3):489-98. doi: 10.1002/cncr.22806. PMID 17592827
- [Background] Kurian AW, Thompson RN, Gaw AF, Arai S, Ortiz R, Garber AM. A cost-effectiveness analysis of adjuvant trastuzumab regimens in early HER2/neu-positive breast cancer. J Clin Oncol. 2007 Feb 20;25(6):634-41. doi: 10.1200/JCO.2006.06.3081. PMID 17308268
- [Background] Liberato NL, Marchetti M, Barosi G. Cost effectiveness of adjuvant trastuzumab in human epidermal growth factor receptor 2-positive breast cancer. J Clin Oncol. 2007 Feb 20;25(6):625-33. doi: 10.1200/JCO.2006.06.4220. PMID 17308267
- [Background] Perez E, Romond E, Suman V, et al.: Updated results of the combined analysis of NCCTG N9831 and NSABP B-31 adjuvant chemotherapy with/without trastuzumab in patiens with HER2-positive breast cancer. [Abstract] J Clin Oncol 25 (Suppl 18): 512, 6s, 2007.
- [Background] Telli ML, Hunt SA, Carlson RW, Guardino AE. Trastuzumab-related cardiotoxicity: calling into question the concept of reversibility. J Clin Oncol. 2007 Aug 10;25(23):3525-33. doi: 10.1200/JCO.2007.11.0106. PMID 17687157
- [Background] Baselga J, Perez EA, Pienkowski T, Bell R. Adjuvant trastuzumab: a milestone in the treatment of HER-2-positive early breast cancer. Oncologist. 2006;11 Suppl 1:4-12. doi: 10.1634/theoncologist.11-90001-4. PMID 16971734
- [Background] Gupta AK, Mekan SF, Eckman MH: Trastuzumab for all? A decision analysis examining tradeoffs between efficacy and cardiac toxicity of adjuvant therapy in HER2 positive breast cancer. [Abstract] J Clin Oncol 24 (Suppl 18): A-6022, 306s, 2006.
- [Background] Burstein HJ. The distinctive nature of HER2-positive breast cancers. N Engl J Med. 2005 Oct 20;353(16):1652-4. doi: 10.1056/NEJMp058197. No abstract available. PMID 16236735
- [Background] Hortobagyi GN. Trastuzumab in the treatment of breast cancer. N Engl J Med. 2005 Oct 20;353(16):1734-6. doi: 10.1056/NEJMe058196. No abstract available. PMID 16236745
- [Background] Tan-Chiu E, Piccart M. Moving forward: Herceptin in the adjuvant setting. Oncology. 2002;63 Suppl 1:57-63. doi: 10.1159/000066201. PMID 12422056
- [Background] Costa RB, Kurra G, Greenberg L, Geyer CE. Efficacy and cardiac safety of adjuvant trastuzumab-based chemotherapy regimens for HER2-positive early breast cancer. Ann Oncol. 2010 Nov;21(11):2153-2160. doi: 10.1093/annonc/mdq096. Epub 2010 Mar 29. PMID 20351072
- [Result] Rastogi P, Jeong J, Geyer CE, et al.: Five year update of cardiac dysfunction on NSABP B-31, a randomized trial of sequential doxorubicin/cyclophosphamide (AC)→paclitaxel (T) vs. AC→T with trastuzumab(H). [Abstract] J Clin Oncol 25 (Suppl 18): A-LBA513, 2007.
- [Result] Geyer CE, Bryant JL, Romond EH, et al.: Update of cardiac dysfunction on NSABP B-31, a randomized trial of sequential doxorubicin/cyclophosphamide (AC)→paclitaxel (T) vs. AC→T with trastuzumab (H). [Abstract] J Clin Oncol 24 (Suppl 18): A-581, 2006.
- [Result] Kim C, Bryant J, Horne Z, et al.: Trastuzumab sensitivity of breast cancer with co-amplification of HER2 and cMYC suggests pro-apoptotic function of dysregulated cMYC in vivo. [Abstract] Breast Cancer Research and Treatment 94 (Suppl 1): A-46, 2005.
- [Result] Tan-Chiu E, Yothers G, Romond E, Geyer CE Jr, Ewer M, Keefe D, Shannon RP, Swain SM, Brown A, Fehrenbacher L, Vogel VG, Seay TE, Rastogi P, Mamounas EP, Wolmark N, Bryant J. Assessment of cardiac dysfunction in a randomized trial comparing doxorubicin and cyclophosphamide followed by paclitaxel, with or without trastuzumab as adjuvant therapy in node-positive, human epidermal growth factor receptor 2-overexpressing breast cancer: NSABP B-31. J Clin Oncol. 2005 Nov 1;23(31):7811-9. doi: 10.1200/JCO.2005.02.4091. PMID 16258083
- [Result] Geyer CE Jr, Bryant J, Romond E: Cardiac safety analysis of the first stage of NSABP B-31, a randomized trial comparing the safety and efficacy of adriamycin® and cyclophosphamide (AC) followed by taxol® to that of AC followed by taxol® plus herceptin® in patients (Pts) with operable, node-positive (N+), HER-2 overexpressing breast cancer (HER2+BC). [Abstract] Breast Cancer Res Treat 82 (Suppl 1): A-23, S13, 2003.
- [Result] Paik S, Bryant J, Tan-Chiu E, Romond E, Hiller W, Park K, Brown A, Yothers G, Anderson S, Smith R, Wickerham DL, Wolmark N. Real-world performance of HER2 testing--National Surgical Adjuvant Breast and Bowel Project experience. J Natl Cancer Inst. 2002 Jun 5;94(11):852-4. doi: 10.1093/jnci/94.11.852. PMID 12048273
- [Result] Romond EH, Perez EA, Bryant J, Suman VJ, Geyer CE Jr, Davidson NE, Tan-Chiu E, Martino S, Paik S, Kaufman PA, Swain SM, Pisansky TM, Fehrenbacher L, Kutteh LA, Vogel VG, Visscher DW, Yothers G, Jenkins RB, Brown AM, Dakhil SR, Mamounas EP, Lingle WL, Klein PM, Ingle JN, Wolmark N. Trastuzumab plus adjuvant chemotherapy for operable HER2-positive breast cancer. N Engl J Med. 2005 Oct 20;353(16):1673-84. doi: 10.1056/NEJMoa052122. PMID 16236738
- [Result] Perez EA, Romond EH, Suman VJ, Jeong JH, Davidson NE, Geyer CE Jr, Martino S, Mamounas EP, Kaufman PA, Wolmark N. Four-year follow-up of trastuzumab plus adjuvant chemotherapy for operable human epidermal growth factor receptor 2-positive breast cancer: joint analysis of data from NCCTG N9831 and NSABP B-31. J Clin Oncol. 2011 Sep 1;29(25):3366-73. doi: 10.1200/JCO.2011.35.0868. Epub 2011 Jul 18. PMID 21768458
- [Derived] Chumsri S, Pai T, Ma Y, Li Z, Gil A, Moreno-Aspitia A, Colon-Otero G, Pogue-Geile KL, Rasgoti P, Paik S, Perez EA, Thompson EA. Clinical Treatment Score Post-5 Years (CTS5) and Late Recurrence Risk in Hormone Receptor-Positive, HER2-Positive Breast Cancer. J Natl Compr Canc Netw. 2024 Aug 26;22(7):463-468. doi: 10.6004/jnccn.2024.7015. PMID 39191270
- [Derived] Chumsri S, Li Z, Serie DJ, Mashadi-Hossein A, Colon-Otero G, Song N, Pogue-Geile KL, Gavin PG, Paik S, Moreno-Aspitia A, Perez EA, Thompson EA. Incidence of Late Relapses in Patients With HER2-Positive Breast Cancer Receiving Adjuvant Trastuzumab: Combined Analysis of NCCTG N9831 (Alliance) and NRG Oncology/NSABP B-31. J Clin Oncol. 2019 Dec 10;37(35):3425-3435. doi: 10.1200/JCO.19.00443. Epub 2019 Oct 17. PMID 31622131
- [Derived] Chumsri S, Serie DJ, Li Z, Pogue-Geile KL, Soyano-Muller AE, Mashadi-Hossein A, Warren S, Lou Y, Colon-Otero G, Knutson KL, Perez EA, Moreno-Aspitia A, Thompson EA. Effects of Age and Immune Landscape on Outcome in HER2-Positive Breast Cancer in the NCCTG N9831 (Alliance) and NSABP B-31 (NRG) Trials. Clin Cancer Res. 2019 Jul 15;25(14):4422-4430. doi: 10.1158/1078-0432.CCR-18-2206. Epub 2019 Feb 26. PMID 30808774
- [Derived] Gavin PG, Song N, Kim SR, Lipchik C, Johnson NL, Bandos H, Finnigan M, Rastogi P, Fehrenbacher L, Mamounas EP, Swain SM, Wickerham DL, Geyer CE Jr, Jeong JH, Costantino JP, Wolmark N, Paik S, Pogue-Geile KL. Association of Polymorphisms in FCGR2A and FCGR3A With Degree of Trastuzumab Benefit in the Adjuvant Treatment of ERBB2/HER2-Positive Breast Cancer: Analysis of the NSABP B-31 Trial. JAMA Oncol. 2017 Mar 1;3(3):335-341. doi: 10.1001/jamaoncol.2016.4884. PMID 27812689
- [Derived] O'Sullivan CC, Bradbury I, Campbell C, Spielmann M, Perez EA, Joensuu H, Costantino JP, Delaloge S, Rastogi P, Zardavas D, Ballman KV, Holmes E, de Azambuja E, Piccart-Gebhart M, Zujewski JA, Gelber RD. Efficacy of Adjuvant Trastuzumab for Patients With Human Epidermal Growth Factor Receptor 2-Positive Early Breast Cancer and Tumors </= 2 cm: A Meta-Analysis of the Randomized Trastuzumab Trials. J Clin Oncol. 2015 Aug 20;33(24):2600-8. doi: 10.1200/JCO.2015.60.8620. Epub 2015 Jun 22. PMID 26101239
- [Derived] Perez EA, Romond EH, Suman VJ, Jeong JH, Sledge G, Geyer CE Jr, Martino S, Rastogi P, Gralow J, Swain SM, Winer EP, Colon-Otero G, Davidson NE, Mamounas E, Zujewski JA, Wolmark N. Trastuzumab plus adjuvant chemotherapy for human epidermal growth factor receptor 2-positive breast cancer: planned joint analysis of overall survival from NSABP B-31 and NCCTG N9831. J Clin Oncol. 2014 Nov 20;32(33):3744-52. doi: 10.1200/JCO.2014.55.5730. Epub 2014 Oct 20. PMID 25332249
- [Derived] Romond EH, Jeong JH, Rastogi P, Swain SM, Geyer CE Jr, Ewer MS, Rathi V, Fehrenbacher L, Brufsky A, Azar CA, Flynn PJ, Zapas JL, Polikoff J, Gross HM, Biggs DD, Atkins JN, Tan-Chiu E, Zheng P, Yothers G, Mamounas EP, Wolmark N. Seven-year follow-up assessment of cardiac function in NSABP B-31, a randomized trial comparing doxorubicin and cyclophosphamide followed by paclitaxel (ACP) with ACP plus trastuzumab as adjuvant therapy for patients with node-positive, human epidermal growth factor receptor 2-positive breast cancer. J Clin Oncol. 2012 Nov 1;30(31):3792-9. doi: 10.1200/JCO.2011.40.0010. Epub 2012 Sep 17. PMID 22987084